CLINICAL TRIAL: NCT05480839
Title: A Comparison of Patient Perceptions Undergoing Manual Immediately Sequential Bilateral Cataract Surgery (M-ISBCS) vs Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery (ReLA-ISBCS)
Brief Title: Manual Immediately Sequential Bilateral Cataract Surgery (M-ISBCS) vs Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery (ReLA-ISBCS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UptownEye2
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: MCS vs ReLACS; Pain Perception Postoperative; Early Anesthesia vs Standard Anesthesia; Immediately Sequential Bilateral Cataract Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual Immediately Sequential Bilateral Cataract Surgery (MCS) (Experimental)
  Interventions: Procedure: M-IBCS
- Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery (ReLA-ISBCS) Early (Experimental)
  Interventions: Procedure: ReLA-IBCS Early
- Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery (ReLA-ISBCS) Standard (Experimental)
  Interventions: Procedure: ReLA-ISBCS

INTERVENTIONS:
Procedure: M-IBCS — Manual Cataract Surgery - Phacoemulsification: removal of the eye lens and insertion of an intraocular lens implant
  Arms: Manual Immediately Sequential Bilateral Cataract Surgery (MCS)
Procedure: ReLA-IBCS Early — Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery - ReLA-IBSCS with early administration of anesthesia
  Arms: Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery (ReLA-ISBCS) Early
Procedure: ReLA-ISBCS — Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery - ReLA-IBSCS with standard administration of anesthesia
  Arms: Refractive Laser-Assisted Immediately Sequential Bilateral Cataract Surgery (ReLA-ISBCS) Standard

SUMMARY:
The focus of this study is to assess the differences in patient perceptions of pain undergoing cataract surgery by using the Refractive Laser-Assisted Cataract Surgery (ReLACS) technique compared to the standard Manual Cataract Surgery (MCS) technique using an immediately sequential bilateral approach. This study also aims to further explore difference in patients' perceptions of pain depending on timing of neurolept anesthesia in the ReLACS technique. The importance of this study is appreciated patient perception of pain during ReLACS, which is an emerging technique for cataract surgery and has been sparsely reported on to date. This investigation will include the analysis of various surgical, ocular, medical, and psychosocial metrics of patients undergoing both ReLACS and MCS at Uptown Eye specialist.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uncomplicated cataract surgery with either surgical technique (M-ISBCS or ReLA-ISBCS)
* Patients who require surgery in both eyes by the same surgeon
* Able to understand English and complete a pain assessment (NRS)

Exclusion Criteria:

* Deafness or communication disorder, known Dementia, Severe COPD/Asthma (severe lung disorder), Severe OSA, Psychiatric or Anxiety conditions, involuntary movement disorders, allergy to the anesthesia, any conditions requiring intraoperative iris manipulation, any prior ocular surgery
* Pre-existing chronic eye pain or uveitis, or complicated cataracts (dislocation, zonulopathy)
* Pre-existing uncontrolled glaucoma/high IOP
* Intraoperative complications or non-routine cataracts (eg. Sutures, excessive time of surgery)
* Any patient who requires Deep Sedation (Propofol), GA or preOP Ativan
* Patients under 40, severe obesity (BMI >35)
* Chronic pain/narcotics/recreational or medical marijuana

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain Perception between Manual Immediately Sequential Bilateral Cataract Surgery (M-ISBCS) and Refractive Laser-Assisted Immediately Sequential Cataract Surgery (ReLA-ISCS) | 1 year
  Pain perceptions of patients undergoing M-IBCS vs ReLA-ISBCS will be measured using the Numerical Rating Scale (NRS) with pain ratings from 0 to 10.

SECONDARY OUTCOMES:
Effects of Early vs Standard administration of topical neurolept anesthesia on pain perception | 1 Year
  Pain perceptions of patients undergoing ReLA-ISBCS Early vs ReLA-ISBCS Standard will be measured using the Numerical Rating Scale (NRS) with pain ratings from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Uptown Eye Specialist, Brampton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No